CLINICAL TRIAL: NCT06155032
Title: Study of Rescue Endovascular Therapy for Progressive Acute Mild Ischemic Stroke With Large Vascular Occlusion--- A Multi-centered, Prospective, Open-label, Blind Endpoint, Randomized Controlled Trial (RESCUE END-LOW)
Brief Title: Rescue Endovascular Therapy for Progressive Acute Mild Ischemic Stroke With Large Vascular Occlusion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Wannan Medical College (Other)
Collaborators: The First Affiliated Hospital of Anhui Medical University (Other); Xiangtan Central Hospital (Other); The First Affiliated Hospital of Hainan Medical University (Other Government); Huang Shan People's Hospital (Other); Fuyang people's hospital (Other); Linyi People's Hospital (Other); Jiujiang No.1 People's Hospital (Other); Taihe Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 20230004
Record Dates: First submitted 2023-11-17; First posted 2023-12-04 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Stroke, Ischemic; Cerebrovascular; Disorder, Occlusive
Keywords: endovascular therapy; mild stroke; neurological deterioration
MeSH Terms: conditions — Ischemic Stroke; Bites and Stings

STUDY DESIGN:
Intervention Model Description: Drug: Best medical management Procedure: Endovascular therapy
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endovascular therapy (Experimental): Patients in this group will receive best medical management plus EVT including mechanical thrombectomy, aspiration thrombectomy, intra-arterial thrombolysis, angioplasty or stenting.
  In the procedure, the methods including mechanical thrombectomy, aspiration thrombectomy, intra-arterial thrombolysis, angioplasty and stenting can be used according to the local interventionalists' choice. Mechanical thrombectomy or aspiration thrombectomy will be recommended as the primary treatment.
  Interventions: Procedure: Endovascular therapy
- Best medical management (Active Comparator): Patients in this group will receive best medical management alone. All the patients enrolled received standard guideline-directed medical therapy including: monitor vital signs, management of blood pressure, glucose and lipids, antithrombotic (antiplatelet or anticoagulant therapy determined by treating physician) therapy if appropriate.
  Interventions: Procedure: Endovascular therapy; Drug: Best medical management

INTERVENTIONS:
Procedure: Endovascular therapy — Patients in this group will receive best medical management plus EVT including mechanical thrombectomy, aspiration thrombectomy, intra-arterial thrombolysis, angioplasty or stenting.
  In the procedure, the methods including mechanical thrombectomy, aspiration thrombectomy, intra-arterial thrombolysis, angioplasty and stenting can be used according to the local interventionalists' choice. Mechanical thrombectomy or aspiration thrombectomy will be recommended as the primary treatment.
  Other Names: EVT group
Drug: Best medical management — All the patients enrolled received standard guideline-directed medical therapy including: monitor vital signs, management of blood pressure, glucose and lipids, antithrombotic (antiplatelet or anticoagulant therapy determined by treating physician) therapy if appropriate
  Other Names: Best medical management group
  Arms: Best medical management

SUMMARY:
Endovascular therapy (EVT) added on best medical management is currently recommended in acute large vascular occlusion (LVO) stroke patients with National Institutes of Health Stroke Scale (NIHSS) score >5. Thus, a sizeable fraction of patients with a minor stroke that do not undergo cerebrovascular screening may experience an early neurological deterioration (END) due to LVO, possibly leading to poor long-term functional outcome. However, whether these patients may still benefit from a rescue EVT is unknown, especially in a late window (>24 hours). In this study, the investigators assume that best medical management plus EVT might be superior than best medical management alone in a late window for minor stroke patients who have experienced an LVO and END. The primary objective of the study was to establish the safety and efficacy of EVT in a late window for minor stroke patients in the anterior circulation who experienced an LVO and END.

DETAILED DESCRIPTION:
The RESCUE END-LOW is a multicentered, prospective, randomized, open-label, blinded end-point (PROBE) study. A total of approximately 272 patients (age ≥ 18 years) in a late window (>24 hours) with a minor stroke (NIHSS <6) who experienced an END and the imaging evidence of an occlusion of the Internal Carotid Artery (ICA) terminus and/or Middle Cerebral Artery Main Stem (MCA M1) segment will be enrolled. Patients fulfilling all of the inclusion criteria and none of the exclusion criteria will be randomized 1:1 into two groups after offering informed content. One group will receive best medical management alone the other group will receive best medical management plus EVT including mechanical thrombectomy, aspiration thrombectomy, intra-arterial thrombolysis, angioplasty or stenting. The primary objective is to establish the efficacy of EVT in a late window for patients with LVO and a minor stroke who have experienced an END. The study consists of seven visits including the day of randomization, 24 hours after randomization, 48 hours, 72 hours, 7 days or discharge, and 30 and 90 days. Demographic information, symptoms and signs, laboratory test, neuro-imaging assessment neurological function rating scale will be recorded during the program. The primary endpoint is the rate of modified Rankin's scale (mRS) 0-2 at 90 days. The trial is anticipated to last from December 2023 to December 2025 with 272 subjects recruited form about 30 centers in China. All the related investigative organization and individuals will obey the Declaration of Helsinki and Chinese Good Clinical Practice standard. A Data and Safety Monitoring Board (DSMB) will regularly monitor safety during the study. The trial has been approved by Institutional Review Board (IRB) and Ethics Committee (EC) in Yijishan Hospital, Wannan Medical College.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria：

* Age ≥ 18 years；
* Presenting with symptoms consistent with an AIS and the initial NIHSS score <6 points；
* Symptom progression within 7 days of first onset；
* Randomization can be finished > 24 hours of stroke onset (stroke onset time is defined as last known well time)；
* Symptom progression to randomization time ≤ 24 hours；
* NIHSS score before randomization ≥ 6 points；
* Informed consent signed.

Specific Neuroimaging Inclusion Criteria

* CTA or MRA proved occlusion of Internal Carotid Artery (ICA) terminal or M1 segment of Middle Cerebral Artery;
* The progression of symptoms is caused by the recurrence of cerebrovascular diseases in the same vascular region, or the pathogenesis is caused by reduced blood flow perfusion;
* NCCT ASPECTS before randomization ≥ 6
* CTP or MRP assessment shows low perfusion in the target vessel area, and meets the following criteria: core infarction volume is less than 50ml, mismatch rate is greater than or equal to 1.8, and mismatch volume is greater than 15ml.

Exclusion Criteria:

* Pre-stroke mRS score >1;
* Imaging confirms the progression of symptoms caused by intracranial hemorrhage, brain edema, or other clear causes;
* The target vessel may have factors that may prevent it from completing endovascular treatment, such as a diameter less than 1.5mm, a tortuous vascular pathway, difficulty in reaching the target position with instruments, or difficulty in recovery;
* Severe stenosis or occlusion of multiple blood vessels;
* Combined with untreated intracranial aneurysms, intracranial tumors (excluding small meningiomas), or intracranial vascular malformations;
* Intracranial hemorrhage within 6 months, including cerebral parenchymal hemorrhage, ventricular hemorrhage, and subarachnoid hemorrhage;
* Have had gastrointestinal or urinary system bleeding, acute myocardial infarction, traumatic brain injury, or undergone major surgical procedures within the past month;
* Known hemorrhagic tendency (including but not limited to): Baseline platelet count <40×109/L; on anticoagulant therapy with warfarin and International Normalized Ratio (INR) > 2 (Patients with no history or suspected coagulopathy do not need to wait for laboratory results of INR or APTT prior to enrollment) Severe heart, liver, kidney function damage or other severe late stage diseases of the system;
* Known allergies to treatment related drugs such as iodine contrast agents, etc; Known severe allergy (more than a rash) to contrast media uncontrolled by medications;
* Refractory hypertension (defined as persistent systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg);
* Uncontrolled blood sugar abnormalities (less than 2.8mmol/l or greater than 22.2mmol/l);
* Females who are pregnant, or those of child-bearing potential with positive urine or serum beta Human Chorionic Gonadotropin (HCG) test;
* The expected survival time is less than 1 year (such as complicated with malignant tumor, serious heart and lung diseases, etc.)
* Participation in other interventional randomized clinical trials that may confound outcome assessment of the trial
* Other circumstances that the investigator considers inappropriate for participation in the trial or that may pose significant risks to patients (such as inability to understand and/or follow the study procedures and/or follow up due to mental disorders, cognitive or emotional disorders)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
90-day good clinical outcome | 90±7 days after randomization
  Good clinical outcome defined as a dichotomized mRS 0-2 outcome

SECONDARY OUTCOMES:
Rate of symptomatic intracranial hemorrhage (sICH) per Heidelberg standard | within 24±6 hours after randomization
  Heidelberg standard was defined as new intracranial hemorrhage detected by brain imaging associated with any of the item below:
  4 points total NIHSS at the time of diagnosis compared to immediately before worsening.
  2 point in one NIHSS category. Leading to intubation/hemicraniectomy/ventricular drainage placement or other major medical/surgical intervention.
  Absence of alternative explanation for deterioration.
Neurofunctional deficit defined as modified Rankin Scale (mRS) | 90±7 days after randomization
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6 with "0" being perfect health without symptoms to "6" being death.
  Score 0: No symptoms Score 1: No significant disability. Able to carry out all usual activities, despite some symptoms.
  Score 2: Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  Score 3: Moderate disability. Requires some help, but able to walk unassisted. Score 4: Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  Score 5: Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  Score 6: Dead
90-day clinical outcome | 90±7 days after randomization
  mRS 0-3 outcome
Change of infarct volume from baseline to 7 days | baseline, 7 days after randomization
  The infarct volume is determined on a diffusion-weighted MRI map based on an ADC threshold of less than 620 ×10-6mm2/s or on CTP image with rCBF<30%
All-cause mortality rate | 90±7 days after randomization
  All-cause mortality rate at 90±7 days
Any type of intracranial hemorrhage according to Heidelberg Classification. | within 24±6 hours after randomization
  Any type of intracranial hemorrhage according to Heidelberg Classification.
1 year clinical outcome | 365±15 days after randomization
  mRS 0-2 outcome
1 year clinical outcome | 365±15 days after randomization
  mRS 0-3 outcome

CONTACTS AND LOCATIONS:
Overall Officials: Zhiming Zhou, PhD, Principal Investigator — The First Affiliated Hospital, Yijishan Hospital of Wannan Medical College; Kai Wang, PhD, Principal Investigator — The First Affiliated Hospital of Anhui Medical University
Locations (7):
- China (7):
  - Fuyang People's Hospital, Fuyang, Anhui
  - First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The first Hospital of Anhui University Of Science & Technology, Huainan, Anhui
  - Huangshan City People's Hospital, Huangshan City, Anhui
  - Wan Bei General Hospital of Wanbei Coal power Group, Suzhou, Anhui
  - The First Affiliated Hospital, Yijishan Hospital of Wannan Medical College, Wuhu, Anhui
  - Xiangyang No.1 People's Hospital, Xiangyang, Hubei

IPD SHARING:
Plan to Share IPD: No